CLINICAL TRIAL: NCT01187277
Title: A Randomized Controlled Trial on Hemiplegic Gait Rehabilitation: Robotic Locomotor Training Versus Conventional Training in Subacute Stroke.
Brief Title: Robotic Versus Conventional Training on Hemiplegic Gait.
Acronym: BB200810
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prasat Neurological Institute (Other Government)
Collaborators: Mahidol University (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ratanapat Chanubol, Dr., Prasat Neurological Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BB200810
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; gait training; robot-assisted therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A = conventional therapy means: 50 min individual physiotherapy and 60 min individual occupational therapy per work day (5x per week)for four consecutive weeks
  Interventions: Behavioral: conventional therapy
- Group B (Active Comparator): Group B = conventional therapy plus robot-assisted means: 30 min individual physiotherapy plus 20 min robot-assisted gait training and 60 min individual occupational therapy per work day (5x per week)for four consecutive weeks
  Interventions: Device: conventional plus robotic gait assisted therapy

INTERVENTIONS:
Behavioral: conventional therapy — conventional therapy means: 50 min individual physiotherapy and 60 min individual occupational therapy per work day (5x per week)for four consecutive weeks
  Arms: Group A
Device: conventional plus robotic gait assisted therapy — individual physiotherapy +individual occupational therapy+ robotic gait assisted therapy
  Other Names: Gait trainer GT1
  Arms: Group B

SUMMARY:
The incidence of stroke in the industrial world is still high. Most of the patients are suffering from paresis of the affected side, speech and cognition problems. Modern concepts of motor learning after stroke favouring a task-specific repetitive high-intensity therapy approach to promote motor outcome. In the last couple of years robot-assisted therapy became an important part of modern rehabilitation after stroke. But so far there is no clear evidence that robot assisted therapy in combination with conventional therapy is more effective than conventional therapy alone to promote motor functions after stroke.

ELIGIBILITY:
Inclusion criteria:

* Subacute first-time stroke patients(hemorrhage and ischemic)
* Age 18-80 years.
* Impaired Functional Ambulation Category at initial score 0-2
* Cardiovascular stable
* Given signed inform consent

Exclusion Criteria:

* Unstable general medical condition
* Severe malposition or fixed contracture of joint with an extension deficit of more than 30 degree
* Any functional impairment prior to stroke
* Can not adequately cooperate in training

  * Severe communication problems
  * Severe cognitive - perceptual deficits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories (FAC, 0-5) | 4 weeks
  Description of ambulation level of the individual patient, whether and if, how much support is needed.
Barthel index (BI, 0-100) | 4 weeks
  Assesses independence in activity of daily living

SECONDARY OUTCOMES:
Berg Balance Scale (BBS, 0-56 | 4 weeks
  Assesses balance abilities.
REPAS -Muscle tone (REPAS, 0-52) | 4 weeks
  Sum score to assess muscle tone for the major joints of the upper and lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Ratanapat Chanubol, M.D., Principal Investigator — Rehabilitation department, Prasat Neurological Institute
Locations (1):
- Prasat Neurological Institute, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Schwartz I, Sajin A, Fisher I, Neeb M, Shochina M, Katz-Leurer M, Meiner Z. The effectiveness of locomotor therapy using robotic-assisted gait training in subacute stroke patients: a randomized controlled trial. PM R. 2009 Jun;1(6):516-23. doi: 10.1016/j.pmrj.2009.03.009. PMID 19627940
- [Result] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Result] Hidler J, Nichols D, Pelliccio M, Brady K, Campbell DD, Kahn JH, Hornby TG. Multicenter randomized clinical trial evaluating the effectiveness of the Lokomat in subacute stroke. Neurorehabil Neural Repair. 2009 Jan;23(1):5-13. doi: 10.1177/1545968308326632. PMID 19109447
- [Result] Pohl M, Werner C, Holzgraefe M, Kroczek G, Mehrholz J, Wingendorf I, Hoolig G, Koch R, Hesse S. Repetitive locomotor training and physiotherapy improve walking and basic activities of daily living after stroke: a single-blind, randomized multicentre trial (DEutsche GAngtrainerStudie, DEGAS). Clin Rehabil. 2007 Jan;21(1):17-27. doi: 10.1177/0269215506071281. PMID 17213237